CLINICAL TRIAL: NCT06931301
Title: Effect of Hyperbaric Oxygen Therapy on Osteonecrosis of the Femoral Head When Combined With 3D Navigated Core Decompression With Bone Marrow Aspirate Concentrate
Brief Title: Effect of HBOT on Femoral Head Avascular Necrosis (AVN)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000038319
Record Dates: First submitted 2025-04-08; First posted 2025-04-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Osteonecrosis; Avascular Necrosis
MeSH Terms: conditions — Osteonecrosis | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Participants with femoral head avascular necrosis having core decompression surgery using 3D modeling techniques with autologous bone marrow aspirate concentrate through the Yale Avascular Necrosis and Osteonecrosis Program. Participants will be able to choose which arm they wish to enroll in by participating in shared clinical decision making with the provider.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Hyperbaric Oxygen Therapy- Full Marx Protocol (Experimental): 30 treatments before surgery, and 10 treatments after surgery
  Interventions: Device: Hyperbaric Oxygen Therapy
- Hyperbaric Oxygen Therapy- Reduced Marx Protocol (Experimental): 20 treatments before surgery and 10 treatments after surgery
  Interventions: Device: Hyperbaric Oxygen Therapy
- Control (No Intervention): No hyperbaric oxygen therapy
- HBOT outside Yale (Experimental): The participant is having HBOT sessions at a different location (outside of the Yale New Haven Health system). These treatments will be overseen by the outside facility's HBOT Director and completed according to the Marx protocol . The patient is responsible for picking a site, setting up their intake appointments, and going to the treatments. The patient is also responsible for providing the HBOT site Director with our protocol as well as returning a completed form that indicates that the proper protocol was used.
  Interventions: Device: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — Sechrist Monoplace Hyperbaric Chamber Model 3600, Chamber will be used to supply patients with 100% oxygen to breathe at 2-2.4 ATA (the equivalent of diving to 33 - 45 feet of sea water) for two hours, 5 treatments per week
  Arms: HBOT outside Yale; Hyperbaric Oxygen Therapy- Full Marx Protocol; Hyperbaric Oxygen Therapy- Reduced Marx Protocol

SUMMARY:
The primary objective of this study is to determine whether the Hyperbaric Oxygen Therapy (HBOT) conducted under the Marx Protocol improves pain outcomes when combined with core decompression with autologous bone marrow aspirate concentrate to treat patients with femoral head avascular necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Diagnosed with femoral head avascular necrosis
* Enrolled into Yale Avascular Necrosis Program
* Avascular necrosis lesion is classified as ARCO I or ARCO II by Investigator
* Surgical Candidate for Core Decompression using 3D image guidance with bone marrow aspirate concentrate

Exclusion Criteria:

* Hip has already collapsed due to severe avascular necrosis (ARCO III or ARCO IV)
* Medical comorbidities that prevent them from being a surgical candidate (example: obesity)
* Absolute contraindications to HBOT, including severe decompensated cardiac failure or lung disease putting them at high risk for pneumothorax
* Pregnant
* Prisoner
* Does not sign Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2035-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Change in Pain scores measured with the Visual Analog Scale (VAS). | baseline, after every 5 treatments of HBOT treatment, 6 weeks, 4.5 months, 9 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  Participants will be asked to mark a point on a 100 mm horizontal line that represents the intensity of their pain. This line has two endpoints: 0: No pain and 10: Worst possible pain imaginable. The distance from the "0" to the mark is measured in millimeters with the resulting number (0-10) being the VAS pain score.

SECONDARY OUTCOMES:
Change in Pain interference PROMIS questionnaire scores | baseline, after every 5 treatments of HBOT treatment, 6 weeks, 4.5 months, 9 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  The PROMIS Pain Interference measures the self-reported consequences of pain on a person's life. Total score range 40 to 80 with higher scores indicating worse outcomes.
Change in Physical function/mobility PROMIS questionnaire scores | baseline, after every 5 treatments of HBOT treatment, 6 weeks, 4.5 months, 9 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  PROMIS Physical Function measures self-reported capability of physical activities. Scores range from 80-20. A lower T-score represents a worse physical function.
Change in Oxford Hip Scores (OHS) | baseline, after every 5 treatments of HBOT treatment, 6 weeks, 4.5 months, 9 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  OHS is an assessment of 12 items of patient-reported outcomes to assess pain and function after hip replacement surgery. Total score range 0 to 48 with higher scores indicating better outcomes.
Change in ARCO classification | baseline, 6 weeks, 4.5 months, 9 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  Number of Participants that had a change in ARCO 2019 classification using x-rays of hip to determine classification.

CONTACTS AND LOCATIONS:
Overall Officials: Rummana Aslam, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health System, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.yalemedicine.org/departments/avascular-necrosis-and-osteonecrosis-program